CLINICAL TRIAL: NCT02160288
Title: Effects of Type A Botulinum Toxin in Obstructed Defecation Syndrome: a Phase II Randomized, Parallel-Group, Triple-Blind, Placebo-Controlled Trial
Brief Title: Effects of Botox in Obstructed Defecation Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low recruitment
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Liliana Bordeianou, Assistant Professor of Surgery, Division of General and Gastrointestinal Surgery, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MGH2014-P-000406
Record Dates: First submitted 2014-06-03; First posted 2014-06-10 (Estimated); Results first posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Obstructed Defecation Syndrome (ODS)
Keywords: Botox; Obstructed Defecation Syndrome; ODS; Outlet-Type Constipation; injection
MeSH Terms: interventions — Botulinum Toxins, Type A; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botulinum Toxin-A (Active Comparator): Patients will receive Botulinum Toxin-A (Botox) injected in the puborectalis muscle and external anal sphincter. We will use 100 units of Botox, a dose with a good safety profile that has been proven to work in previous studies performed in adults.
  Interventions: Drug: Botulinum Toxin-A
- Normal saline (Placebo Comparator): Patients will receive normal saline (placebo) injected in the puborectalis muscle and external anal sphincter.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Botulinum Toxin-A — 100 Units diluted in a 5 cc syringe at a concentration of 20U/mL
  Other Names: Botox
  Arms: Botulinum Toxin-A
Drug: Normal Saline — Dispensed in a 5 cc syringe
  Other Names: 0.9% Sodium Chloride
  Arms: Normal saline

SUMMARY:
The purpose of this study is to determine if Botulinum Toxin-A (Botox) injection will improve symptoms of constipation in obstructed defecation syndrome (ODS).

DETAILED DESCRIPTION:
Constipation represents one of the five most common physician diagnoses for gut disorders. Obstructed defecation syndrome (ODS) is an under-treated condition which accounts for 30%- 50% of all patients with constipation and it is more common as people age. ODS is due to the abnormal contraction of the puborectalis muscle (a muscle around the anus that should relax during defecation).

Biofeedback therapy and medical management are the standards of care for ODS. Typically patients are first managed with dietary modifications (fiber supplementation, increased fluids) and medication (laxatives, enemas). If constipation is not improved, they will undergo biofeedback, which lasts from 3-8 sessions on average. Biofeedback acts on the cause of ODS and it has good short-term success, but around 50%-70% of treated patients re-experience constipation after one year. The main drawbacks of biofeedback for ODS are the facts that it is expensive, time-consuming, available in few select-centers and its success depends very much on the provider. Biofeedback is delivered in multiple 1-hour clinic sessions, so many patients don't finish all recommended sessions and their constipation may recur faster.

Botox also acts on the cause of ODS and was shown to improve constipation within 1-3 weeks after the injection. Botox is delivered as a one-time injection in the puborectalis muscle and external anal sphincter (the muscle right around the anus). The injection can be performed in the clinic under local anesthesia, and the patient goes home afterwards. Currently, Botox is used for treatment of patients who fail biofeedback and medical management, to avoid the options of last resort (resection of the colon with stoma). To this day, no adequately designed study has confirmed that Botox is indeed superior to placebo (normal saline) for the treatment of ODS. The results from this study will provide valuable data on the ability of Botox to improve symptoms of constipation and the duration of its effect. This project has the potential to increase the availability of effective treatments for ODS.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 years or older of all races and backgrounds
* Competent to give informed consent
* Meet the Rome III diagnostic criteria for functional constipation
* Inability to relax the puborectalis muscle at electromyography
* Altomare Obstructed Defecation Syndrome score of 15 points or above
* Failure of treatment with 2 conservative measures which may be as follows:

  * 1 laxative (osmotic or stimulant) for 2 weeks
  * 1 fiber supplement for one month
  * And/or trial of biofeedback for at least 4 sessions

Exclusion Criteria:

* Previous treatment with Botox (possible antibodies)
* Known hypersensitivity to any of the components of the toxin
* Medication regimen includes narcotics
* Previous radiation therapy to the anal canal and rectum
* Prior proctectomy
* Presence of unhealed and symptomatic anal fissure
* Presence of anal pain
* Presence of fecal incontinence
* Presence of full thickness rectal prolapse
* Presence of internal sphincter myopathy
* Inflammatory bowel disease or proctitis
* Pregnancy or breast-feeding
* Subject is currently enrolled/ just finished participating in a clinical trial in which the intervention/ its carry-over effect may interact with the intervention in this trial

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2019-06-11 (Actual); Study Completion 2019-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Liliana Bordeianou, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Shaheen NJ, Hansen RA, Morgan DR, Gangarosa LM, Ringel Y, Thiny MT, Russo MW, Sandler RS. The burden of gastrointestinal and liver diseases, 2006. Am J Gastroenterol. 2006 Sep;101(9):2128-38. doi: 10.1111/j.1572-0241.2006.00723.x. Epub 2006 Jul 18. PMID 16848807
- [Background] Suares NC, Ford AC. Prevalence of, and risk factors for, chronic idiopathic constipation in the community: systematic review and meta-analysis. Am J Gastroenterol. 2011 Sep;106(9):1582-91; quiz 1581, 1592. doi: 10.1038/ajg.2011.164. Epub 2011 May 24. PMID 21606976
- [Background] American Gastroenterological Association; Bharucha AE, Dorn SD, Lembo A, Pressman A. American Gastroenterological Association medical position statement on constipation. Gastroenterology. 2013 Jan;144(1):211-7. doi: 10.1053/j.gastro.2012.10.029. No abstract available. PMID 23261064
- [Background] Maria G, Cadeddu F, Brandara F, Marniga G, Brisinda G. Experience with type A botulinum toxin for treatment of outlet-type constipation. Am J Gastroenterol. 2006 Nov;101(11):2570-5. doi: 10.1111/j.1572-0241.2006.00791.x. Epub 2006 Oct 4. PMID 17029615

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Botulinum Toxin-A | Normal Saline
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: We were unable to recruit more than one patient to the study so it was closed
Groups:
- Total: Total of all reporting groups
Arm/Group | Botulinum Toxin-A | Normal Saline | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 0 | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 0 | 1
ODS score [Number; unit: units on a scale] | 20 |  | 20

OUTCOME MEASURES:

1. Primary Outcome: Changes in the Altomare Obstructed Defecation Syndrome- Score (ODS-S) and Patient Assessment of Constipation- Quality of Life Score (PAC-QoL)
Description: The primary outcome measure will be the change from baseline in the sum of ODS-S and PAC-QoL at 1 month after the Botox injection.
  This measures the symptomatic improvement in ODS. ODS (altomare obstructed defecation syndrome score) scores range from 0 (minimum) to 31 (maximum) where 31 is the most severe (worse outcome) and 0 is no symptoms (better outcome).
  The scale for PAC-QoL (Patient Assessment of Constipation- Quality of life score) is a minimum of 0 and a maximum of 112 where 0 is highest quality of life (better outcome) and 112 is lowest quality of life (worse outcome)
  Larger number for change would suggest a better outcome
Time Frame: Baseline, 1 month after injection
Population: since there was only one participant, analysis of the data is limited
Measure: Number; unit: change in score on a scale
Arm/Group | Botulinum Toxin-A | Normal Saline
Number analyzed (Participants) | 1 | 0
change in score on a scale | 3 |

2. Secondary Outcome: Changes in the Altomare ODS Score (ODS-S)
Description: The scale title is obstructed defecation score, the minimum value is 0 and the maximum value is 31 for the ODS score. This measures the symptomatic improvement in ODS. ODS scores range from 0-31 where 31 is the most severe and 0 is no symptoms. A higher score would suggest a better outcome.
Time Frame: Assessed at baseline, 1, 3, 6 and 12 months after injection and value compared from baseline to 12 months
Population: since there was only one participant, analysis of the data is limited
Measure: Number; unit: score on a scale
Arm/Group | Botulinum Toxin-A | Normal Saline
Number analyzed (Participants) | 1 | 0
score on a scale | 18 |

3. Secondary Outcome: Changes in the Patient Assessment of Constipation- Quality of Life Score (PAC-QoL)
Description: PAC-QoL is Patient Assessment of Constipation- Quality of Life Score. The scale for PAC-QoL is 0 minimum score to 112 maximum score where 0 is highest quality of life (better outcome) and 112 is lowest quality of life (worse outcome). Since we are looking for a change in score, the minimum change would be 0 and the maximum change would be 112. A higher change would suggest a better outcome.
Time Frame: Assessed at baseline, 1, 3, 6 and 12 months after injection and value compared from baseline to 12 months
Population: since there was only one participant, analysis of the data is limited
Measure: Number; unit: change in score on a scale
Arm/Group | Botulinum Toxin-A | Normal Saline
Number analyzed (Participants) | 1 | 0
change in score on a scale | 21 |

4. Secondary Outcome: Changes in Health-Related Quality of Life
Description: Medical outcomes survey short form (SF-36 version 1) will be used to measure changes in the health-related quality of life.This is a measure of efficacy. The score ranges from 0-100 where 0 is maximum impact on health and 100 is no impact on health
Time Frame: Baseline, 1, 3, 6 and 12 months after injection and value compared from baseline to 12 months
Population: since there was only one participant, analysis of the data is limited
Measure: Number; unit: change in score on a scale
Arm/Group | Botulinum Toxin-A | Normal Saline
Number analyzed (Participants) | 1 | 0
change in score on a scale | 1 |

5. Secondary Outcome: Changes in Cleveland Clinic Fecal Incontinence Score (CCFI)
Description: This is a measure of Botox-specific adverse events. The score is a total of answers of questions. The score range is 0-20 where 0 is perfect incontinence and 20 is complete incontinence.
Time Frame: Assessed at baseline, 1, 3, 6 and 12 months after injection and value compared from baseline to 12 months
Population: since there was only one participant, analysis of the data is limited
Measure: Number; unit: change in score on a scale
Arm/Group | Botulinum Toxin-A | Normal Saline
Number analyzed (Participants) | 1 | 0
change in score on a scale | 2 |

6. Secondary Outcome: Changes in Fecal Incontinence Quality of Life Scale (FIQoL)
Description: This is a measure of Botox-specific adverse events. This fecal incontinence quality of life scale (FIQoL) scale ranges from 4 as the minimum and 20 as maximum. lower score indicates lower quality of life (worse outcome) and higher score has better quality of life (better outcome).
Time Frame: Assessed at baseline, 1, 3, 6 and 12 months after injection and value compared from baseline to 12 months
Population: since there was only one participant, analysis of the data is limited
Measure: Number; unit: change in score on a scale
Arm/Group | Botulinum Toxin-A | Normal Saline
Number analyzed (Participants) | 1 | 0
change in score on a scale | 18 |

7. Secondary Outcome: Relaxation of Puborectalis With Push Measured by EMG
Description: This is a measure of efficacy.
Time Frame: Baseline, 1 month follow-up visit
Population: since there was only one participant, analysis of the data is limited
Measure: Number; unit: participants
Arm/Group | Botulinum Toxin-A | Normal Saline
Number analyzed (Participants) | 1 | 0
participants | 0 |

8. Secondary Outcome: Success of Balloon Expulsion Test
Description: This is a measure of efficacy.
Time Frame: Baseline, 1 month follow-up visit
Population: since there was only one participant, analysis of the data is limited
Measure: Count of Participants; unit: Participants
Arm/Group | Botulinum Toxin-A | Normal Saline
Number analyzed (Participants) | 1 | 0
Participants | 1 |

9. Secondary Outcome: Change in Anal Sphincter Function
Description: The changes in anal sphincter function will be assessed by anorectal manometry. This test will measure the resting sphincter pressure, maximal resting anal pressure, maximum squeeze pressure. The change in anal sphincter function is a measure of treatment efficacy. The minimum score for resting sphincter pressure is 0 and the maximum is 200. The minimum squeeze pressure is 10 and the maximum is 200. The lower score is suggested of decreased tone and worse outcome, where high scores may suggest worse outcome in terms of sphincter function.
Time Frame: Baseline, 1 month follow-up visit
Population: since there was only one participant, analysis of the data is limited
Measure: Number; unit: change of score
Arm/Group | Botulinum Toxin-A | Normal Saline
Number analyzed (Participants) | 1 | 0
change of score | 56.3 |

10. Secondary Outcome: Change in Defecation Index
Description: The defecation index=maximum rectal pressure during attempted defecation/minimum anal residual pressure during attempted defecation. This is calculated based on measurements obtained from anorectal manometry and is a measure of treatment efficacy. Scores can change from 0 (meaning no change- least effective) to 1 meaning that the change shows complete relaxation with defecation.
Time Frame: Baseline, 1 month follow-up visit
Population: since there was only one participant, analysis of the data is limited
Measure: Number; unit: change in score on a scale
Arm/Group | Botulinum Toxin-A | Normal Saline
Number analyzed (Participants) | 1 | 0
change in score on a scale | 0 |

ADVERSE EVENTS:
Time Frame: 3 months
Description: since there were no patients recruited in the saline arm, there is no risk for serious adverse event or mortality
Arm/Group | Botulinum Toxin-A | Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-08-18): https://cdn.clinicaltrials.gov/large-docs/88/NCT02160288/Prot_SAP_000.pdf
  • Informed Consent Form (2016-11-28): https://cdn.clinicaltrials.gov/large-docs/88/NCT02160288/ICF_001.pdf